CLINICAL TRIAL: NCT04277988
Title: A Comparison of the Ultrasound Measured Posterior Longitudinal Ligament Length in Parturients in the Standard Sitting and Crossed Leg Positions: an Observational Study
Brief Title: Effect of Crossed Legged Position on Ultrasound Measured Posterior Longitudinal Ligament Length in Parturients.
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 107570
Record Dates: First submitted 2017-08-24; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2015-12

CONDITIONS: Pregnancy
Keywords: Maternal Analgesia; Ultrasonography Lumbar Spine
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Crossed leg position: Patients in this group will be randomly allocated to sit in crossed leg position first.Ultrasonography will be performed in this position to measure the best visualized length of posterior longitudinal ligament, ligamentum flavum and interlaminar distance at L3-4 lumbar level as by Operator 1 . These measurements will be recorded by Operator 2 using intrinsic caliper software.Operator 1 will not be told the measurements.
  Interventions: Device: Ultrasonography
- Standard Sitting position: Patients in this group will be randomly allocated to sit in standard position first.Ultrasonography will be performed in this position to measure the best visualized length of posterior longitudinal ligament, ligamentum flavum and interlaminar distance at L3-4 lumbar level as by Operator 1 . These measurements will be recorded by Operator 2 using intrinsic caliper software.Operator 1 will not be told the measurements.
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Length of Posterior Longitudianl Ligament, Ligamentum Flavum and Interlaminar distance visible in paramedian longitudinal view during lumbar spine ultrasonography in cross legged position will be compared to standard sitting position.

SUMMARY:
To investigate if sitting in flexed cross legged position for neuraxial techniques in term pregnant patients widens the size of the ultrasound acoustic window as measured by the visualized posterior longitudinal ligament length, during lumbar spine ultrasonography using longitudinal paramedian view, in comparison to the standard sitting flexed position.

DETAILED DESCRIPTION:
This is a prospective observational study involving a total of 30 healthy term gestation pregnant patients with singleton fetuses.Patients will be randomly allocated to sit crossed leg or in standard position first. Using ultrasonography, the acoustic window for lumbar spinal anesthesia at L3-4 will be evaluated in both traditional sitting and crossed leg positions. Ultrasonography will be performed sequentially to measure the best visualized length of posterior longitudinal ligament,ligamentum flavum and interlaminar distance in the paramedian view.The scanned image will be saved to be remeasured by a third observer. Patients will be asked to score their comfort level while sitting in both positions.

ELIGIBILITY:
Inclusion Criteria:

Term gestation Singleton pregnancy 18 years or older Patients having elective cesarean delivery or induction of labor or in early labor

Exclusion Criteria:

* Allergy to ultrasound jelly
* Spinal Deformities/Previous spinal surgery
* No contraindication to neuraxial placement
* Any fetal concerns
* Morbid obesity
* Language barrier

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients at term in the Labour and Delivery Suite, as well as those booked for elective cesarean sections who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
PLL length | Up to Five minutes
  Length of the Paravertebral Longitudinal Ligament, as measured by the intrinsic ultrasound caliber tool in mm.

SECONDARY OUTCOMES:
LF length | Up to Five minutes
  Length of the Ligamentum Flavum as measured by the intrinsic ultrasound caliber tool in mm.
ILD length | Up to Five minutes
  Length of the interlaminar distance, as measured by the intrinsic ultrasound caliber tool in mm.
Patient Comfort | Up to 5 minutes
  Patient comfort level measured on a 1-5 Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Indu Singh, FRCPC, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: Undecided